CLINICAL TRIAL: NCT07191912
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Long-Term Clinical Benefit of Govorestat in Patients With Charcot-Marie-Tooth-Sorbitol Dehydrogenase Deficiency (CMT-SORD)
Brief Title: Confirmatory Study of Govorestat in CMT-SORD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-007-1020
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Charcot-Marie-Tooth Disease With Sorbitol Dehydrogenase Deficiency (CMT-SORD)

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Govorestat and its matching placebo will have the same presentation, the same aspect and taste in order to be indistinguishable, and they will be supplied and used in the same conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Govorestat (Active Comparator): Govorestat is an aldose reductase inhibitor
  Interventions: Drug: Govorestat
- Placebo (Placebo Comparator): Non-active control
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Govorestat — Govorestat will be provided as a liquid suspension (200mg/mL) for weight-based administration and administered orally at 20 mg/kg QD (every 24 hours)
  Other Names: AT-007
  Arms: Govorestat
Drug: Placebo Control — Placebo will also be provided as a matching liquid suspension to be taken orally QD
  Arms: Placebo

SUMMARY:
This study is designed to assess the long-term efficacy and clinical benefit of AT-007 in patients with CMT-SORD. This randomized, double-blind study will assess the effect of govorestat compared to placebo in patients with CMT-SORD for up to 36 months.

DETAILED DESCRIPTION:
This international, multi-center, randomized, double-blinded, placebo-controlled, phase 3 study is designed to assess the efficacy and clinical benefit of long-term govorestat administration to patients with CMT-SORD utilizing functional, patient-reported, and clinical outcomes measures including the CMT-HI, 10MWRT, dorsiflexion, the CMT-FOM, and CMT-related lower extremity muscle MRI parameters along with the long-term effect of govorestat on whole blood sorbitol. Long-term safety of govorestat will also be evaluated.

Patients (16 to 65 years old) with CMT-SORD will be stratified according to their sex (male vs female) and age before randomization in a 2:1 ratio to govorestat 20 mg/kg once daily (QD) or placebo.

There will be a pre-planned Interim Analysis at 2 years (Month 24). If clinical benefit is determined to be met with the Interim Analysis, the study will end and not continue to 3 years.

The study will be conducted at up to 16 sites worldwide. Approximately 155 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
* Male and non-pregnant, non-lactating female patients between the ages of 16 and 65 years, inclusive.
* Females must be of non-childbearing potential (defined as surgically sterile [i.e., had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy ≥6 months prior to the first dose of study drug] or postmenopausal for ≥1 year [confirmatory follicle stimulating hormone or FSH test results required] prior to the first dose of study drug) or agree to use a highly effective form of birth control from Screening until 30 days after the last dose of study drug.
* Males must be unable to procreate (defined as surgically sterile [i.e., had a vasectomy ≥6 months prior to Screening]) or must agree to use a highly effective form of birth control from Screening through 105 days (sum of 5 half-lives and 90 days interval as per CTFG guidelines) after the last dose of study drug.
* Clinical diagnosis of Charcot-Marie-Tooth Type 2 (CMT2) or distal Hereditary Motor Neuropathy (dHMN) due to CMT-SORD confirmed by medical record or written communication by health care professional, elevated blood sorbitol level (>10,000 ng/mL), and SORD gene analysis report indicating at least one pathogenic mutation.
* Patient may be on concomitant medications and dietary supplements; however, they must be on stable doses for at least 1 month prior to Screening and throughout the study. In addition, all over-the-counter (OTC) and/or prescription medications must be reviewed and approved by the Investigator.

Exclusion Criteria:

* Absence of force generated in one or both feet with dorsiflexion (value of 0 Newton).
* History or presence of clinically significant hematopoietic, renal, hepatic, endocrine (e.g. diabetes), metabolic, pulmonary, neurological (e.g. other neuropathy, myopathy or neuromuscular disorder), psychiatric, cardiovascular, immunological, dermatological, or gastrointestinal diseases that are - a priori - altering the proper evaluation of the safety and efficacy of govorestat; conditions capable of altering the absorption, metabolism, or elimination of drugs; or conditions that constitute a risk factor when taking the study drug and/or impact the conduct or results of the study.
* Body Mass Index (BMI) >35 kg/m2.
* Clinically relevant underweight, weight loss suggestive of a pathology unrelated to CMT-SORD, or BMI < 17.5 kg/m2.
* Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at Screening or previous treatment for hepatitis B, hepatitis C, or HIV infection.
* Individuals who smoke or use tobacco or nicotine-containing products.
* Pregnant, lactating, or not using/not willing to use appropriate means of contraception.
* Any prior history of substance abuse (including alcohol) or treatment for such.
* Positive urine drug screen (UDS) for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates) or cotinine.
* Non-ambulatory disability.
* Lower limb surgery such as bilateral ankle stabilization or contracture release in the past 5 years.
* Impaired renal function or estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m2. Note: The eGFR is an estimation of renal function, and the ultimate decision of whether a patient has normal renal function (and can be included in the study) is at the discretion of the Investigator, assuming there are no safety concerns. Also, because eGFR can vary from day to day based on outside factors, patients can be re screened for eGFR multiple times to understand the renal function of the patient.
* Hemoglobin (Hgb) < 10.0 g/dL at Screening.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin (except in case of Gilbert's syndrome) > 1.5 x upper limit of normal (ULN) at Screening.
* Urinary albumin-to-creatinine ratio (UACR) > 30 mg/g at Screening in the presence of elevated creatinine (>2X ULN).
* History or presence of cardiovascular disorders including myocardial infarction, stroke, uncontrolled hypertension (sitting blood pressure ≥140/90 mmHg), left ventricular (LV) hypertrophy, atrial fibrillation, or valvular heart disease considered clinically significant by the Investigator and/or Sponsor medical representative.
* Abnormal findings on the Screening 12-lead ECG, such as ST/T wave changes, pathological Q wave changes, or any rhythm other than normal sinus rhythm considered clinically significant by the Investigator and/or Sponsor medical representative.
* Evidence of significant active hematological disease and/or cumulative blood donation of 1 unit (500 mL) or more including blood drawn during clinical studies in the last 3 months.
* History of significant drug allergy or drug hypersensitivity.
* Investigators, site personnel directly affiliated with this study, and their immediate families (defined as a spouse, parent, child, or sibling, whether biological or legally adopted).
* Any other condition that, in the opinion of the Investigator, precludes the patient from following and completing the protocol.
* A clinically significant abnormal finding on the physical exam, medical history or clinical laboratory results at Screening.
* A significantly abnormal diet (per Investigator judgment) during the 4 weeks preceding the first dose of study drug.
* Participation in another clinical study of a different investigational product within 30 days prior to the first dose of study drug.
* Use of any OTC medication (including nutritional or dietary supplements, herbal preparations, or vitamins) ≤7 days prior to the first dose of study drug until the last dose of study drug without evaluation and approval by the Investigator.
* Use of any prescription medication, except those allowed per protocol, from 30 days prior to the first dose of study drug until the last dose of study drug without evaluation and approval by the Investigator.
* Treatment with any sensitive substrates of Breast Cancer Resistance Protein (BCRP) or potent inhibitors of BCRP.
* Treatment with any sensitive substrates of cytochrome P450 3A4 (CYP3A4), CYP2B6, CYP2C19, or CYP1A2.
* Treatment with any sensitive substrates of Organic Anion Transporter (OAT)1 and OAT3. Treatment with any drugs potentially associated with transaminase elevations. Potentially nephrotoxic drugs are prohibited.
* Consumption of beverages or foods that contain alcohol, high levels of sorbitol, grapefruit, poppy seeds, broccoli, brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study drug through the last dose of study drug. Patients will be instructed not to consume any of the above products; however, allowance for sporadic consumption may be evaluated and approved by the Investigator based on the potential for interaction with the study drug. Not more than half cup of coffee per day should be consumed.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Charcot-Marie-Tooth, Health Index (CMT-HI) Total Score | From enrollment to the end of treatment at 36 months
  The CMT-HI is a disease-specific, validated, patient-reported measure that is largely focused on functional items in addition to activities of daily living and emotional well-being. The CMT-HI was designed to assess specific impact of CMT disease and to remove redundancy.

SECONDARY OUTCOMES:
10-meter walk-run test (10MWRT) | From enrollment to the end of treatment at 36 months
  The 10MWRT is a timed functional test used to measure walking or running speed over 10 meters by the study population
Dorsiflexion | From enrollment to the end of treatment at 36 months
  Maximum isometric dorsiflexion force measured in Newtons using a calibrated dynamometer in a standardized position; higher values indicate greater dorsiflexion strength.
Charcot-Marie-Tooth, Health Index (CMT-HI) Sub-Domain Scores | From enrollment to the end of treatment at 36 months
  The CMT-HI is a disease-specific, validated, patient-reported measure that is largely focused on functional items in addition to activities of daily living and emotional well-being. The CMT-HI was designed to assess specific impact of CMT disease and to remove redundancy. The CMT-HI has 18 sub-domains, each of which will be evaluated separately.
Charcot Marie Tooth Functional Outcome Measure (CMT-FOM) | From enrollment to the end of treatment at 36 months
  The CMT-FOM is a performance-based measure that assesses the functional ability of patients with CMT. There are 5 domains (strength, upper limb function, lower limb function, balance, and motility) that are assessed by 13 test items specifically selected to ensure functional/patient-relevance, reliability/validity, and responsiveness to change. Total and sub-domain scores of the CMT-FOM, will be evaluated to detect change over time.
Muscle Magnetic Resonance Imaging (MRI) | From enrollment to the end of treatment at 36 months
  Patients will undergo MRI of their legs to evaluate the fat deposition and the muscle size, both CMT-related parameters of disease progression.
Whole blood sorbitol levels | From enrollment to the end of treatment at 36 months
  Patients with CMT-SORD develop extremely high sorbitol levels in cells and tissues, as aldose reductase converts glucose to sorbitol which then cannot be converted into fructose by SORD. Sorbitol is known to be toxic to many cell types. Prior studies have shown a correlation of sorbitol levels with different clinical outcomes in CMT-SORD. We will evaluate the effect of govorestat on whole blood sorbitol levels over time.
Plasma drug concentration | From enrollment through Month 3
  Plasma drug concentration samples will be obtained pre-dose (within 60 minutes) and at 2, 4, 6, 8 hours after the dose.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Clinic for Special Children, Gordonville, Pennsylvania
- Sydney Childrens, Sydney, Australia
- France (2):
  - CHU La Timone, Marseille
  - Institut de Myologie, Paris
- Germany (3):
  - Uniklinik of the RWTH Aachen University, Aachen
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Medicine Gottingen (UMG), Göttingen
- Carlo Besta Neurological Institute, Milan, Italy
- Spain (2):
  - Vall d'Hebron Institut de Recerca (VHIR), Barcelona
  - La Fe University and Polytechnic Hospital, Valencia
- Turkey (Türkiye) (2):
  - Koç University Hospital, Istanbul
  - Istanbul University, Istanbul

IPD SHARING:
Plan to Share IPD: No